CLINICAL TRIAL: NCT03362567
Title: Comparative Effects of Sustained Natural Apophyseal Glides and Mechanical Cervical Traction in the Management of Cervical Radiculopathy
Brief Title: Sustained Natural Apophyseal Glides and Mechanical Cervical Traction in the Management of Cervical Radiculopathy
Acronym: SNAG&MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Dr and Senior Lecturer, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPHOAU/12/673
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy; Sustained Natural Apophyseal Glides; Mechanical Cervical Traction; Pain Intensity; Neck Disability
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Intervention Model Description: The study involved 47 patients with cervical radiculopathy which were purposively recruited from the Physiotherapy Department Outpatient Clinic of Usmanu Danfodio University Teaching Hospital, Sokoto for the study. Subjects were randomly allocated to Sustained Natural Apophyseal Glides (SNAGS)and Mechanical Cervical Traction (MCT) group. All the subjects were treated using cryotherapy for seven minutes. Subjects in SNAGS group were then treated with sustained natural apophyseal glides, twice weekly for six weeks while subjects in MCT received mechanical cervical traction, for 15 minutes each session twice in a week for six weeks. Visual analogue scale, neck disability index questionnaires and inclinometer were used to assess pain intensity, disability and cervical range of motion respectively at the beginning, 3rd and 6th week of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAGS Group (Experimental): Subjects in SNAGS group were treated with application of sustained natural apophyseal glides, twice weekly for six weeks
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Mechanical Cervical Traction
- MCT Group (Experimental): subjects in MCT received mechanical cervical traction, for 15 minutes each session twice in a week for six weeks
  Interventions: Other: Sustained Natural Apophyseal Glides; Other: Mechanical Cervical Traction

INTERVENTIONS:
Other: Sustained Natural Apophyseal Glides — Subjects in SNAGS group were treated with sustained natural apophyseal glides, twice weekly for six weeks
  Other Names: SNAGS
Other: Mechanical Cervical Traction — subjects in MCT received mechanical cervical traction, for 15 minutes each session twice in a week for six weeks
  Other Names: MCT

SUMMARY:
Sustained natural apophyseal glides (SNAGS), is a form of manual therapy, involved a combination of a sustained facet glide with active motion, followed by overpressure. Natural apophseal glides (NAGS), a modification of SNAGS, involves a mid to end-range facet joint mobilisation applied anterocranially or posterioanteriorly along the plane of treatment, combined with a small amount of manual traction which increases movement within the spine, and decreases symptomatic pain . A study reported that Natural Apophyseal Glides (NAGS) and Sustained Natural Apophyseal Glides (SNAGS) demonstrated significant effects in reducing pain and disability in subjects with chronic neck pain . This technique, SNAGS, is however an evolving manual therapy techniques which its effectiveness has not been thoroughly investigated in cervical radiculopathy treatment raised author's curiosity to compare and document efficacy of SNAGS with cervical traction in Nigeria since comparative studies evaluating SNAGS and manual cervical traction relative efficacies among Nigerians are yet to be documented if at all available. Consequently, the quest is to look for a quicker and a better way of relieving cervical radiculopathy in this environment . The more reason why we have to compare it with a conventional mechanical traction.

DETAILED DESCRIPTION:
This is a Quasi experimental study. Participants will be patients with radiculopathy receiving treatment at the Usman Danfodio University Teaching Hospital Sokoto Nigeria. Ethical approval will be obtained from Institute of Public Health of the Obafemi Awolowo University Ile-Ife, Nigeria, and a copy will be taken to the site of the study. The purpose and protocol for the study will be explained to the participants, after their informed consent have been obtained. The sample size will be determined using N= 4σ2 (Zcrit+Zpwr)2/ D2 where N is the total sample size, σ is the assumed SD of each group (assumed to be equal for the groups), which is assumed to be 16.63 from previous study; Zcrit is the standard normal deviate corresponding to the selected significance criterion, i.e 0.05(95% = 1,960), Zpwr is the standard normal deviate corresponding to the selected statistical power (i.e. 0.80 = 0.842), and D is the minimum expected difference among the three means, and D =18 from a previous study. Therefore, N obtained will be 41.22. Fifty two participants are proposed for this study (making 26 participants for each group) in order to give room for attrition. The 52 participants will be allocated to two groups (Groups A and B) using permuted block randomization. Subjects in group A will receive (i) Sustained Natural Apophyzeal Glides: Each subject in this group will be in sitting position facing the wall bar. The therapist will place on thumb reinforced over the spinous process of the implicated cervical vertebra. The therapist will then push upon the implicated spinous process. The pressure will be sustained for 60 seconds. Six repetitions will be carried out and maintained on each visit twice in a week for 6 weeks. Subjects in group B will receive over -the -door mechanical cervical traction in sitting position using position 10% of each patient's body weight for 15 minutes on each visit, twice in a week for 6 weeks. Pain intensity will be measured using visual analogue scale, cervical range of motions will be measured using inclinometer, functional disabilities will be measured using neck disabilities index questionnaires. The out come measures will be applied three times: pre-treatment, 3rd week and 6th week within the treatment period. The data obtained will be analysed using descriptive and inferential statistics.

ELIGIBILITY:
Inclusion Criteria: Subjects diagnosed with neck pain of mechanical origin of not less than 3 months. Subjects without pathology affecting the neck and upper limb(s).

-

Exclusion Criteria:(i) Participants with history of vertebro-basilary artery insufficiency. Patient with history of cervical surgery or arthroplasty

-

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 6 weeks
  Visual analogue scale is a scale with 10 points indicating the severity of pain. o indicate no pain and 10 indicate excruciating pain. 5 indicate moderate pain. Patient is asked to point to the scale indicating the perception of his or her pain intensity

SECONDARY OUTCOMES:
Neck disability index | 6 weeks
  It has 10 sections with 5 questions on each section asking patient on what he can do. Patient circles one choice that is most appropriate to him. These are added together and percentage are found. If 9 are filled out of 10 it will be 9 multiplied by 5 making 45. The total score divided by 45 multiply by 100 will be the percentage of disability. If the percentage is high, the disability is high and if the percentage is low the disability is low

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo, Phd, Principal Investigator — Obafemi Awolowo University

REFERENCES:
- [Background] Ali A, Shakil-Ur-Rehman S, Sibtain F. The efficacy of Sustained Natural Apophyseal Glides with and without Isometric Exercise Training in Non-specific Neck Pain. Pak J Med Sci. 2014 Jul;30(4):872-4. PMID 25097535